CLINICAL TRIAL: NCT04166604
Title: LONsurf and G-CSF Use: Being On A Right Dose-intensity to Optimize Treatment Efficacy
Acronym: LONGBOARD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LONGBOARD C19-01
Record Dates: First submitted 2019-11-04; First posted 2019-11-18 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: trifluridine/ tipiracil; G-CSF; neutropenia
MeSH Terms: conditions — Colorectal Neoplasms; Neutropenia | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: It was planned to include 250 patients in a prospective cohort, to obtained 89 patients in the phase II (experience a grade 3-4 neutropenia)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- trifluridine/tipiracil (Experimental): 35mg/m² BID (PER OS) (one cycle every 4 weeks)
  Interventions: Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — After morning and evening meal
  Days 1 through 5: 35mg/m2 (twice daily)
  Days 6 through 7: recovery
  Days 8 through 12: 35mg/m2 (twice daily)
  Day 13 through 28: recovery
  Other Names: Lonsurf

SUMMARY:
Prospective cohort of patients treated with trifluridine/tipiracil, maximal sample size 250 patients. It is expected, that 89 patients will experience a grade 3-4 neutropenia and will be included in the phase II.

DETAILED DESCRIPTION:
Trifluridine/tipiracil has demonstrated its efficacy in patients with metastatic colorectal cancer (mCRC) resistant to standard drugs (fluoropyrimidine, oxaliplatin, irinotecan, bevacizumab, and panitumumab or cetuximab in case of RAS wild-type tumors). This treatment has a marketing authorization.

Neutropenia is a classic complication of cytotoxic treatments. Febrile neutropenia are associated with a mortality rate of 9.5% and a hospitalization of 6 days in median. Recent meta-analyses have reported that the use of granulocyte-colony stimulating factor (GCSF) allows to maintain the dose-intensity of cytotoxic treatment and was associated with a better overall survival (OS).

There is currently no clear recommendation for the use of G-CSF with trifluridine/tipiracil.

Unpublished analyses that various clinical parameters may be associated with the risk of neutropenia: age ≥ 65 years, female sex, level of leukocytes at baseline, and time of initial diagnostic to randomization ≥ 36 months.These data are too preliminary to allow proposing a G-CSF primary prophylaxis in a defined subgroup of patients. However, a secondary prophylaxis based on the administration of G-CSF seems efficient, with a prescription from day 14 to day 18.

The aim of this phase II study is to assess the efficacy of the secondary prophylaxis with G-CSF in case of first episode of grade 3-4 neutropenia in the aim to maintain the optimal dose intensity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent,
2. Patients willing and able to comply with protocol requirements,
3. Histologically proven colorectal adenocarcinoma,
4. Stage IV disease,
5. Have life expectancy of at least 6 months,
6. Previous chemotherapy regimens with each of the following agents: fluoropyrimidine, oxaliplatin, irinotecan, anti-vascular endothelial growth factor (VEGF) therapy (bevacizumab, aflibercept), and anti-epidermal growth factor receptor (EGFR) therapy (cetuximab or panitumumab for tumors with wild-type RAS and/or BRAF wild type),
7. At least one measurable or evaluable lesion as assessed by computed tomography (CT)-scan or magnetic resonance imaging (MRI) according to RECIST v1.1,
8. Age ≥ 18 years,
9. ECOG PS 0-1,
10. Adequate hematologic function: neutrophils > 1.5 x 109 /L; platelets > 100 x 109 /L; hemoglobin ≥ 9 g/dL,
11. Calculated creatinine clearance ≥ 30 mL/min,
12. Adequate liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit normal ULN;

    ≤ 5 x ULN in case of liver metastasis), total bilirubin ≤ 1.5 x ULN (< 2 x ULN if hyperbilirubinemia is due to Gilbert's syndrome), albumin ≥ 25 g/L,
13. Baseline evaluations: clinical and blood evaluations no more than 14 days prior to inclusion and start of trifluridine/tipiracil, Tumor assessment (CT-scan or MRI, evaluation of non-measurable lesions) no more than 21 days prior to inclusion and start of trifluridine/tipiracil,
14. Female patients must be surgically sterile, or be postmenopausal, or must commit to using reliable and appropriate methods of contraception during the study (must have a negative pregnancy test within 7 days prior to enrollment) and during at least 6 months after the end of the last dose of study treatment (when applicable). All female patients with reproductive potential must have a negative pregnancy test (β-HCG) within 72 hours prior to starting trifluridine/tipiracil treatment. Breastfeeding is not allowed. Male patients must agree to use effective contraception in addition to having their partner use a contraceptive method as well during the trial and during at least 6 months after the end of the study treatment,
15. Registration with the French National Health Care System or PUMA (Protection Universelle MAladie).

Exclusion Criteria:

1. Medical history or evidence of CNS metastasis upon physical examination, unless adequately treated (e.g. non-irradiated CNS metastasis, seizure not controlled with standard medical therapy, patients are stable without evidence of progression for at least 28 days prior to the first dose of treatment),
2. Local or locally advanced disease (stage I to III),
3. Treatment with warfarin,
4. Uncontrolled hypercalcemia,
5. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
6. Known complete dihydropyrimidine dehydrogenase (DPD) deficiency,
7. Treatment with any other investigational medicinal product within 28 days prior to study entry,
8. Symptomatic carcinomatosis with occlusive symptoms or ascites requiring paracentesis,
9. Other serious and uncontrolled non-malignant disease (e.g. active infection requiring systemic therapy, coronary stenting or myocardial infarction, or stroke in the past 6 months),
10. HIV-infected patients or otherwise known to be HIV-positive,
11. Untreated hepatitis B or C,
12. Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for > 5 years,
13. Concomitant administration of prophylactic phenytoin and live attenuated virus vaccine such as yellow fever vaccine 28 days prior to the first dose of treatment.
14. Patient under guardianship, curatorship or under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Rate of patients free of trifluridine/tipiracil dose reduction or postponement of cycles of > 7 days at 6 months or at progression or death or stop of treatment for another cause than neutropenia if observed in 6 months. | At 6 months
  To assess, in mCRC patients treated with trifluridine/tipiracil after the introduction of G-CSF in a secondary prevention attempt, the rate of patients free of trifluridine/tipiracil dose reduction or postponement of cycles of > 7 days at 6 months from G-CSF first intake date or at progression or death or stop of treatment for another cause than neutropenia if observed in the 6 months.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 30 months
  OS - defined as the time from study enrollment to death (from any cause) or to the last date the patients was known to be alive
Progression free survival (PFS) | Up to 30 months
  PFS - defined as the time (in months) from study enrollment until objective PD or death from any cause. If the patient dies before reaching PD, the date of death is considered as the date that PD was reached. For patients that had not reached PD at the time of the analysis, and for patients for whom the PD date is unknown, PFS is censored at the date of patient's final assessment prior to data cut-off.
Objective response rate (ORR) | Up to 30 months
  ORR - defined as proportion of patients with reduction in tumor burden of predefined amount. It refers to the number of patients with CR, PR according to RECIST v1.1
Disease control rate (DCR) | Up to 30 months
  The disease control rate (DCR) is defined as the proportion of patients in whom the best overall response is determined as complete response, partial response or stable disease
Safety descriptive analysis | Up to 30 months
  Patients will be assessed for AEs throughout the study at every visit during treatment. Investigators using the NCI-CTCAE version 5.0 will grade the severity of AEs.
The rate of dose reductions | Up to 30 months
  Number of patients for whom a dose reduction was required and the reasons for dose reduction,
Clinical or biological factors at baseline associated with the occurrence of grade 3-4 neutropenia | Up to 30 months
  Identification of clinical and biological factors at baseline associated with the occurrence of grade 3-4 neutropenia in the whole cohort and design of predictive model of neutropenia occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jean Baptiste BACHET, MD, Principal Investigator — Hôpital Pitié Salpêtrière
Locations (22):
- France (22):
  - CHU Amiens, Amiens
  - Institut de cancérologie de l'Ouest, Angers
  - CHRU Jean Minjoz, Besançon
  - centre Pierre Curie, Beuvry
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre hospitalier de Chauny, Chauny
  - Polyclinique Sainte Côme, Compiègne
  - Clinique de Flandre, Coudekerque-Branche
  - Hôpital Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital Franco-Britannique, Levallois-Perret
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Européen, Marseille
  - Hôpital Layne, Mont-de-Marsan
  - Hôpital Nord Franche Comté, Montbéliard
  - Groupe Hospitalier Pitié Sapêtrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Haut Lévêque, Pessac
  - CHU Poitiers, Poitiers
  - CHU Robert Debré, Reims